CLINICAL TRIAL: NCT03598504
Title: Closed Loop Control of Vibration for Muscular Spasms After Human Spinal Cord Injury: Efficacy and Mechanism
Brief Title: Vibration for Muscle Spasms After Spinal Cord Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Monica Perez, Scientific Chair Arms + Hands AbilityLab, Shirley Ryan AbilityLab
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STU00209996; 1R01NS100810-01A1 (NIH)
Record Dates: First submitted 2018-07-13; First posted 2018-07-26 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Spinal Cord Injuries
Keywords: SCI; Spasms; Vibration
MeSH Terms: conditions — Spinal Cord Injuries; Spasm

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Clinical measures of spasticity before, during, and after the intervention will be implemented by an evaluator blind to the treatment effects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Controls Group (Active Comparator): 1. A focus group to gather information about the perceptions, opinions, beliefs, and attitudes towards management of muscle spasms by vibration using our portable device, information that will drive design improvement (size, fit, weight).
  Interventions: Device: Wearable EMG/Vibration device
- Spinal Cord Injury Group (Active Comparator): 1a. A focus group to gather information about the perceptions, opinions, beliefs, and attitudes towards management of muscle spasms by vibration using our portable device, information that will drive design improvement (size, fit, weight).
  1b. In the lab, we will trigger spasms in paralyzed leg muscles in one of two common postures (seated, reclined), detect the contractions using electromyography (EMG), and condition alternate spasms with vibration using our custom device. We will examine the vibration parameters that reduce muscle spasms best.
  2. Participants will complete 1 or 2 multi-day experiments. EMG (24-hour) data will be collected at baseline (day 1), during the vibration intervention (day 2), and post intervention (day 3) to examine the acute effects of vibration on muscle spasms
  Interventions: Device: Wearable EMG/Vibration device

INTERVENTIONS:
Device: Wearable EMG/Vibration device — The device is a combination of an EMG recorder/detector and a vibrator

SUMMARY:
This study uses closed-loop control of tendon vibration to implement clinically meaningful management of muscle spasms after spinal cord injury (SCI), and to understand the mechanisms responsible for spasm generation change in response to vibration.

DETAILED DESCRIPTION:
The specific aims of this study are listed below:

1a) Evaluate the ergonomics of the wearable device that will be used to record and detect spasms, then to deliver vibration to tendons to dampen spasms.

1. b) Determine the vibration parameters that best reduce spasms in leg muscles paralyzed by spinal cord injury (SCI) in the laboratory using the wearable device.
2. a) Examine the efficacy of tendon vibration in altering muscle spasms by treating spasms as they occur in real world environments using 24-hour electromyographic (EMG) recordings.

Hypothesis 2a: Achilles tendon vibration will dampen spasms acutely, and may alter their distribution Assess excitatory and/or inhibitory mechanisms that underlie spasms, and changes induced with vibration, by recording physiological, clinical, functional and self-reported measures of different aspects of spasticity, and health-related quality of life, before and after conditioning spasms with vibration. These data will provide insight into the site(s), magnitude, and time-course of changes with vibration; and user perspective on the effects of the therapy.

Achilles tendon vibration will dampen spasms by reconfiguring circuits generating 6-13 Hz shared drive to motoneurons.

ELIGIBILITY:
Inclusion Criteria:

* Male and females between ages 18-85 years of age
* SCI ( ≥1 month of injury)
* ASIA A, B,C and D
* SCI above L5
* Able to perform a visible contraction with dorsiflexor and hip flexor muscles (allowing testing of largely impaired patients)
* Able to ambulate a few steps with or without an assistive device.

Inclusion criteria for healthy controls:

* Male and females between ages 18-85 years
* Able to complete precision grips with both hands
* Able to complete full elbow flexion-extension with both arms.
* Able to walk and complete lower-limb tests with both legs.

Exclusion Criteria:

* Uncontrolled medical problems including pulmonary, cardiovascular or orthopedic disease,
* Any debilitating disease prior to the SCI that caused exercise intolerance
* Premorbid, ongoing major depression or psychosis, altered cognitive status
* History of head injury or stroke,
* Metal plate in skull
* History of seizures
* Receiving drugs acting primarily on the central nervous system, which lower the seizure threshold such as antipsychotic drugs (chlorpromazine, clozapine) or tricyclic antidepressants.
* Pregnant females, and
* Ongoing cord compression or a syrinx in the spinal cord or who suffer from a spinal cord disease such as spinal stenosis, spina bifida or herniated cervical disk.

This information will be obtained by self-report.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2019-07-16 (Actual); Primary Completion 2022-12-15 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in muscle spasms with vibration device | 4 weeks
  Measured by records of EMG from 4 muscles to quantify spasms

SECONDARY OUTCOMES:
Questionnaire | 10 minutes
  Quantitative and qualitative survey for subjects developed to evaluate comfort and user-friendliness of device. The questionnaire includes 11-point scale questions to rate spasms and effect of the device (0 means no effect and 10 means complete satisfaction. Values for each answer will be interpreted separately and a 10 signifies a better outcome); dichotomous (yes/no) questions about the device, where "no" signifies no interruption to their different routines and therefore "no" represents a better outcome; and free-answer questions to collect qualitative data on concerns and recommendations.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Perez, PhD, PT, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States